CLINICAL TRIAL: NCT00447382
Title: A 12-months Multi-national, Multi-centre, Double Blind, Randomised, Parallel Safety and Efficacy Comparison of Insulin Detemir Produced by the Current Process and Insulin Detemir Produced by the NN729 Process in Subjects With Type 1 Diabetes on a Basal-bolus Regimen With Insulin Aspart as the Bolus Insulin
Brief Title: Safety of Insulin Detemir Produced by a New Process as Measured by Antibody Formation in Subjects With Type 1 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EX1729-1778; 2006-004733-15 (EudraCT Number)
Record Dates: First submitted 2007-03-13; First posted 2007-03-14 (Estimated); Results first posted 2011-05-12 (Estimated); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin Detemir; Insulin Aspart

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NN304 (Active Comparator): Individually adjusted dosage of insulin detemir produced by the NN304 process, administered sub-cutaneously (s.c.) 1-2 times daily + Individually adjusted dosage of insulin aspart, administered sub-cutaneously (s.c.) at meals for 52 weeks
  Interventions: Drug: insulin detemir; Drug: insulin aspart
- NN729 (Experimental): Individually adjusted dosage of insulin detemir produced by the NN729 process, administered sub-cutaneously (s.c.) 1-2 times daily + Individually adjusted dosage of insulin aspart, administered sub-cutaneously (s.c.) at meals for 52 weeks
  Interventions: Drug: insulin aspart; Drug: insulin detemir

INTERVENTIONS:
Drug: insulin detemir — NN304 injected s.c. (under the skin). Given as basal insulin.
  Arms: NN304
Drug: insulin aspart — Injected s.c. (under the skin). Given as bolus insulin.
Drug: insulin detemir — NN729 injected s.c. (under the skin). Given as basal insulin
  Arms: NN729

SUMMARY:
The trial was conducted in Germany, The Republic of Macedonia, Russian Federation, Serbia and South Africa. The aim of this trial was to make a safety comparison of insulin detemir produced by a new production method (NN729) with insulin detemir made by the previous production method (NN304). Subjects were treated with NN729 or NN304 for a period of 52 weeks at the same total daily dose and frequency of administration as their own pre-trial basal insulin . During the trial doses were individualised based on subject's plasma glucose measurements.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes for at least 12 months
* Basal-bolus treatment for at least 3 months
* Body Mass Index (BMI) less than or equal to 35.0 kg/m^2
* HbA1c (glycosylated haemoglobin) less than or equal to 12.0%

Exclusion Criteria:

* Known or suspected allergy to trial products or related products
* Pregnancy, breast-feeding or the intention to become pregnant or not using adequate contraceptive measures
* Receipt of any trial drug within 1 month prior to this trial
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation
* Conditions that may interfere with trial participation as judged by Investigator: proliferative retinopathy or maculopathy requiring acute treatment within the last six months, recurrent major hypoglycaemia, impaired hepatic or renal function, cardiac problems, uncontrolled hypertension (treated and untreated)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2007-03; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (5):
- Frankfurt, Germany
- Skopje, North Macedonia
- Moscow, Russia
- Belgrade, Serbia and Montenegro
- Cape Town, Western Cape, South Africa

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty four sites in five countries: Germany (12), The Republic of Macedonia (1), Russian Federation (4), Serbia (3) and South Africa (4)
Pre-assignment Details: Eligible subjects were adults with type 1 diabetes treated with a basal-bolus regimen for at least 3 months prior to the study, who had a BMI (Body Mass Index) no greater than 35.0 kg/m^2 and HbA1c no greater than 12.0%.
Period: Overall Study
Arm/Group | NN304 | NN729
Started | 164 | 166
Completed | 158 | 160
Not Completed | 6 | 6
Not completed — Adverse Event | 1 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Protocol Violation | 2 | 0
Not completed — Unclassified | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NN304 | NN729 | Total
Number analyzed (Participants) | 164 | 166 | 330
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.9 (14.9) | 38.6 (13.6) | 39.3 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 79 | 145
  Male | 98 | 87 | 185
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 152 | 152 | 304
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 9 | 9 | 18
Height [Mean (Standard Deviation); unit: meter] | 1.74 (0.09) | 1.72 (0.1) | 1.73 (0.1)
Body weight [Mean (Standard Deviation); unit: kg] | 77.6 (14.6) | 75.1 (14.9) | 76.4 (14.7)
BMI (Body Mass Index) [Mean (Standard Deviation); unit: kg/m^2] | 25.68 (4.05) | 25.23 (3.59) | 25.45 (3.83)
HbA1c (Glycosylated haemoglobin) [Mean (Standard Deviation); unit: Percent (%) glycosylated haemoglobin] | 7.93 (1.31) | 7.99 (1.38) | 7.96 (1.35)
Diabetes History [Mean (Standard Deviation); unit: years] — Average number of years since diagnosis
  years | 14.48 (11.2) | 13.66 (10.3) | 14.07 (10.8)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Insulin Detemir - Human Insulin Cross-reacting Antibodies
Description: Measured change in concentrations of insulin detemir cross-reacting antibodies and the change ratio from baseline to end of trial was calculated. The unit for measuring antibody levels is %B/T (amount of tracer bound to the antibodies in the precipitate (B) expressed in percentage of the total amount of tracer (T) added to the mixture). The change ratio does not have any unit as it is a ratio.
Time Frame: week 0, week 52
Population: FAS (Full Analysis Set) All randomised subjects exposed to at least one dose of trial product with a post-baseline observation.
Measure: Mean (Standard Error); unit: ratio
Arm/Group | NN304 | NN729
Number analyzed (Participants) | 158 | 152
ratio | 1.81 (0.07) | 1.89 (0.07)
Statistical Analysis 1: Comparison: NN304 vs NN729; Null hypothesis:Treatment with detemir produced with the NN729 process result in a similar change in cross reacting antibody levels as the NN304 process. Alternative hypothesis: change in antibody levels differ after treatment with detemir produced by the two manufacturing processes. The statistical analysis applies to the change from baseline to week 52 which was analysed using ANOVA; Test type: Superiority or Other; p = 0.649, ANOVA; Treatment, previous insulin detemir exposure and country as fixed effects and the baseline value as a covariate. (Log transformed data); Treatment Ratio = 1.04, 95% CI [0.86 to 1.26] — The treatment ratio calculated is the NN729-NN304 ratio for the change from baseline to Week 52. The 95% confidence interval for this ratio was also calculated

2. Secondary Outcome: Hypoglycaemic Episodes
Description: Number of hypoglycaemic episodes from Week 0 to Week 52, defined as major, minor, or symptoms only. Major if unable to treat her/himself. Minor if able to treat her/himself and plasma glucose below 3.1 mmol/L. Symptoms only if able to treat her/himself and no plasma glucose measurement or plasma glucose higher than or equal to 3.1 mmol/L. Hypoglycaemic episodes occurring in the time frame between 23:00 hours (included) and 06:00 hours (excluded) were defined as nocturnal.
Time Frame: Weeks 0-52
Population: All randomised subjects exposed to at least one dose of trial product with a post-baseline observation.
Measure: Number; unit: episodes
Arm/Group | NN304 | NN729
Number analyzed (Participants) | 164 | 166
episodes
  All events - Major | 21 | 21
  All events - Minor | 3215 | 2996
  All events - Symptoms Only | 445 | 318
  Daytime - Major | 9 | 15
  Daytime - Minor | 2741 | 2590
  Daytime - Symptoms Only | 381 | 258
  Nocturnal - Major | 12 | 6
  Nocturnal - Minor | 472 | 404
  Nocturnal - Symptoms Only | 64 | 60
  Unclassified - Minor | 2 | 2

3. Secondary Outcome: Glycaemic Control Parameters (Change in HbA1c)
Description: HbA1c (Glycosylated haemoglobin).
Time Frame: week 0, week 52
Population: All randomised subjects exposed to at least one dose of trial product with a post-baseline observation.
Measure: Mean (Standard Error); unit: Percent (%) glycosylated haemoglobin
Arm/Group | NN304 | NN729
Number analyzed (Participants) | 164 | 165
Percent (%) glycosylated haemoglobin
  Week 52 | 7.88 (0.07) | 7.85 (0.07)
  Change from Baseline to week 52 | -0.08 (0.07) | -0.11 (0.07)
Statistical Analysis 1: Comparison: NN304 vs NN729; The statistical analysis applies to the change from baseline to week 52 which was analysed using ANOVA; Test type: Superiority or Other; p = 0.758, ANOVA; Adjustments: Treatment, previous insulin detemir exposure and country as fixed effects and the baseline value as covariate; Estimated treatment difference = -0.03, 95% CI [-0.21 to 0.15] — The estimated treatment difference calculated is the NN729-NN304 treatment difference for the change from baseline to Week 52. The 95% confidence interval for this difference was also calculated

4. Secondary Outcome: Glycaemic Control Parameters (Change in Fasting Plasma Glucose [FPG])
Time Frame: week 0, week 52
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | NN304 | NN729
Number analyzed (Participants) | 164 | 165
mmol/L
  Week 52 | 9.73 (0.3) | 9.64 (0.3)
  Change from Baseline to week 52 | 0.07 (0.3) | -0.02 (0.3)
Statistical Analysis 1: Comparison: NN304 vs NN729; The statistical analysis applies to the change from baseline to week 52 which was analysed using ANOVA; Test type: Superiority or Other; p = 0.812, ANOVA; [statistical method as in outcome 3, analysis 1]; Estimated treatment difference = -0.1, 95% CI [-0.89 to 0.7] — [estimate comment as in outcome 3, analysis 1]

5. Secondary Outcome: Glycaemic Control Parameters (9-point Self Measured Plasma Glucose [SMPG])
Description: 1. point is Before Breakfast
  2. point is 120 minutes after Breakfast
  3. point is Before Lunch
  4. point is 120 minutes after Lunch
  5. point is Before Dinner
  6. point is 120 minutes after Dinner
  7. point is at Bedtime
  8. point is At 03:00 A.M.
  9. point is Before Breakfast the Following Day
Time Frame: week 0, 26 and 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | NN304 | NN729
Number analyzed (Participants) | 164 | 166
mmol/L
  Baseline 1. point | 8.17 (3.26) | 8.17 (3.56)
  Baseline 2. point | 8.95 (3.86) | 9.03 (3.81)
  Baseline 3. point | 7.66 (3.36) | 7.34 (3.51)
  Baseline 4. point | 8.60 (3.70) | 8.18 (3.74)
  Baseline 5. point | 8.29 (3.37) | 8.16 (3.84)
  Baseline 6. point | 8.43 (3.37) | 8.60 (3.75)
  Baseline 7. point | 8.69 (3.48) | 8.60 (3.70)
  Baseline 8. point | 7.97 (3.51) | 7.72 (3.47)
  Baseline 9. point | 8.05 (3.49) | 7.56 (3.24)
  Week 26 change. 1. point | -0.64 (3.95) | -0.44 (4.38)
  Week 26 change. 2. point | -0.61 (4.43) | -0.61 (4.81)
  Week 26 change. 3. point | -0.49 (3.64) | 0.08 (4.04)
  Week 26 change. 4. point | -0.34 (3.82) | -0.22 (4.27)
  Week 26 change. 5. point | -0.36 (4.22) | -0.00 (4.32)
  Week 26 change. 6. point | -0.35 (4.16) | 0.07 (4.7)
  Week 26 change. 7. point | -0.35 (3.63) | 0.20 (4.37)
  Week 26 change. 8. point | 0.18 (4.05) | 0.08 (4.19)
  Week 26 change. 9. point | -0.64 (4.05) | 0.24 (3.54)
  Week 52 change. 1. point | -0.60 (4.08) | -0.67 (3.85)
  Week 52 change. 2. point | -0.54 (4.80) | -0.99 (4.04)
  Week 52 change. 3. point | -0.36 (3.96) | -0.28 (4.06)
  Week 52 change. 4. point | -0.78 (3.98) | -0.29 (3.93)
  Week 52 change. 5. point | -0.41 (3.80) | -0.59 (4.33)
  Week 52 change. 6. point | -0.31 (4.13) | -0.51 (4.04)
  Week 52 change. 7. point | -0.34 (3.92) | -0.47 (3.68)
  Week 52 change. 8. point | -0.24 (3.59) | -0.31 (3.77)
  Week 52 change. 9. point | -0.44 (4.14) | -0.09 (3.49)

6. Secondary Outcome: Change From Baseline in Detemir Specific Antibodies
Description: Measured change in concentrations of antibody values for insulin detemir specific antibodies and the change ratio from the baseline to end of trial was calculated. The unit for measuring antibody levels is %B/T (amount of tracer bound to the antibodies in the precipitate (B) expressed in percentage of the total amount of tracer (T) added to the mixture). The change ratio does not have any unit as it is a ratio.
Time Frame: Week 0, week 52
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ratio
Arm/Group | NN304 | NN729
Number analyzed (Participants) | 150 | 150
ratio | 1.14 (0.04) | 1.06 (0.04)
Statistical Analysis 1: Comparison: NN304 vs NN729; The statistical analysis applies to the change from baseline to week 52 which was analysed using ANOVA. The analysis was based on an assumption of a log-normal distribution for antibody data and was thus built on log-transformed data; Test type: Superiority or Other; p = 0.15, ANOVA; Adjustments:Treatment, previous insulin detemir exposure and country as fixed effects and the baseline value as a covariate. (Log transformed data); Treatment Ratio = 0.93, 95% CI [0.84 to 1.03] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Change From Baseline in Total Antibodies
Description: Measured change in concentrations of total insulin antibodies values (the sum of insulin detemir specific and insulin detemir - human insulin cross-reacting antibodies) and the change ratio from baseline to end of trial was calculated. The unit for measuring antibody levels is %B/T (amount of tracer bound to the antibodies in the precipitate (B) expressed in percentage of the total amount of tracer (T) added to the mixture). The change ratio does not have any unit as it is a ratio.
Time Frame: Week 0, week 52
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ratio
Arm/Group | NN304 | NN729
Number analyzed (Participants) | 150 | 147
ratio | 1.55 (0.05) | 1.55 (0.05)
Statistical Analysis 1: Comparison: NN304 vs NN729; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.966, ANOVA; Adjustments: Treatment, previous insulin detemir exposure and country as fixed effects and the baseline value as a covariate. (Log transformed data); Treatment Ratio = 1, 95% CI [0.87 to 1.15] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Clinical Laboratory Values (Change in Haematology - Basophilis)
Description: Change from Baseline to Week 52 is calculated from the change in percentage ((Week 52 %) - (Baseline %)) per participant, averaged across all participants.
  Measured in serum at baseline and week 52. Serum samples were analysed at a central laboratory.
Time Frame: week 0, week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent (%) of white blood cells
Arm/Group | NN304 | NN729
Number analyzed (Participants) | 17 | 12
Percent (%) of white blood cells
  Baseline | 0.30 (0.67) | 0.36 (0.50)
  Week 52 | 0.24 (0.56) | 0.33 (0.49)
  Change from Baseline to week 52 | -0.25 (0.50) | 0.00 (0.00)

9. Secondary Outcome: Clinical Laboratory Values (Change in Haematology - Eosinophils)
Description: as for outcome 8
Time Frame: Week 0, week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent (%) of white blood cells
Arm/Group | NN304 | NN729
Number analyzed (Participants) | 10 | 11
Percent (%) of white blood cells
  Baseline | 2.50 (1.27) | 1.82 (1.40)
  Week 52 | 2.47 (2.10) | 2.08 (2.35)
  Change from Baseline to week 52 | -0.25 (2.22) | 0.00 (3.61)

10. Secondary Outcome: Clinical Laboratory Values (Change in Haematology - Haemoglobin)
Description: as for outcome 8
Time Frame: Week 0, week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | NN304 | NN729
Number analyzed (Participants) | 161 | 160
mmol/L
  Baseline | 8.85 (0.92) | 8.80 (0.79)
  Week 52 | 8.54 (0.91) | 8.47 (0.76)
  Change from Baseline to week 52 | -0.30 (0.52) | -0.31 (0.50)

11. Secondary Outcome: Clinical Laboratory Values (Change in Haematology - Lymphocytes)
Description: Change from Baseline to Week 52 is calculated from the change in percentage((Week 52 %) - (Baseline %)) per participant, averaged across all participants.
  Measured in serum at baseline and week 52. Serum samples were analysed at a central laboratory.
Time Frame: Week 0, week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent (%) of white blood cells
Arm/Group | NN304 | NN729
Number analyzed (Participants) | 10 | 11
Percent (%) of white blood cells
  Baseline | 33.80 (6.94) | 37.45 (7.66)
  Week 52 | 28.12 (9.17) | 36.67 (9.30)
  Change from Baseline to week 52 | -3.25 (9.18) | 5.33 (6.66)

12. Secondary Outcome: Clinical Laboratory Values (Change in Haematology - Monocytes)
Description: as for outcome 8
Time Frame: Week 0, week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent (%) of white blood cells
Arm/Group | NN304 | NN729
Number analyzed (Participants) | 4 | 3
Percent (%) of white blood cells
  Baseline | 3.40 (2.17) | 4.00 (2.61)
  Week 52 | 3.59 (2.92) | 3.42 (2.15)
  Change from Baseline to week 52 | -2.50 (1.91) | 0.67 (0.58)

13. Secondary Outcome: Clinical Laboratory Values (Change in Haematology - Neutrophils)
Description: as for outcome 11
Time Frame: Week 0, week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent (%) of white blood cells
Arm/Group | NN304 | NN729
Number analyzed (Participants) | 10 | 11
Percent (%) of white blood cells
  Baseline | 60.00 (7.51) | 56.36 (7.46)
  Week 52 | 65.59 (10.75) | 57.50 (9.60)
  Change from Baseline to week 52 | 6.25 (10.37) | -6.00 (8.66)

14. Secondary Outcome: Clinical Laboratory Values (Change in Haematology - Thrombocytes)
Description: as for outcome 11
Time Frame: Week 0, week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 10^9/L
Arm/Group | NN304 | NN729
Number analyzed (Participants) | 163 | 165
10^9/L
  Baseline | 254.0 (65.5) | 267.1 (59.5)
  Week 52 | 242.2 (58.3) | 247.2 (51.3)
  Change from Baseline to week 52 | -12.8 (38.5) | -18.6 (38.9)

15. Secondary Outcome: Clinical Laboratory Values (Change in Haematology - Leucocytes)
Description: as for outcome 11
Time Frame: Week 0, week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent (%) of white blood cells
Arm/Group | NN304 | NN729
Number analyzed (Participants) | 164 | 166
Percent (%) of white blood cells
  Baseline | 6.22 (1.91) | 6.3 (1.71)
  Week 52 | 6.24 (1.85) | 5.96 (1.55)
  Change from Baseline to week 52 | 0.03 (1.77) | -0.32 (1.69)

16. Secondary Outcome: Clinical Laboratory Values (Change in Biochemistry - Albumin)
Description: as for outcome 11
Time Frame: Week 0, week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | NN304 | NN729
Number analyzed (Participants) | 164 | 166
g/dL
  Baseline | 4.30 (0.23) | 4.27 (0.23)
  Week 52 | 4.28 (0.25) | 4.30 (0.22)
  Change from Baseline to week 52 | -0.02 (0.21) | 0.02 (0.20)

17. Secondary Outcome: Clinical Laboratory Values (Change in Biochemistry - Alanine Aminotransferase [ALAT])
Description: Change from Baseline to Week 52 is calculated from the change in percentage((Week 52 %) - (Baseline %)) per participant, averaged across all participants. Measured in serum at baseline and week 52. Serum samples were analysed at a central laboratory.
  (ALAT = alanine aminotransferase)
Time Frame: Week 0, week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | NN304 | NN729
Number analyzed (Participants) | 164 | 166
U/L
  Baseline | 29.21 (22.12) | 25.98 (13.65)
  Week 52 | 30.72 (25.48) | 27.81 (16.05)
  Change from Baseline to week 52 | 1.34 (17.80) | 1.76 (17.17)

18. Secondary Outcome: Clinical Laboratory Values (Change in Biochemistry - Alkaline Phosphatase [ALP])
Description: Change from Baseline to Week 52 is calculated from the change in percentage((Week 52 %) - (Baseline %)) per participant, averaged across all participants. Measured in serum at baseline and week 52. Serum samples were analysed at a central laboratory.
  (ALP = alkaline phosphatase)
Time Frame: Week 0, week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | NN304 | NN729
Number analyzed (Participants) | 161 | 161
U/L
  Baseline | 75.40 (23.26) | 75.55 (25.30)
  Week 52 | 82.35 (47.20) | 80.42 (23.98)
  Change from Baseline to week 52 | 6.77 (42.36) | 4.53 (15.88)

19. Secondary Outcome: Clinical Laboratory Values (Change in Biochemistry - Creatinine)
Description: as for outcome 11
Time Frame: Week 0, week 52
Population: FAS (Full Analysis Set) All randomised subjects exposed to at least one dose of trial product with a postbaseline observation.
Measure: Mean (Standard Deviation); unit: Umol/L
Arm/Group | NN304 | NN729
Number analyzed (Participants) | 164 | 166
Umol/L
  Baseline | 73.1 (15.4) | 72.3 (31.6)
  Week 52 | 72.5 (16.4) | 73.1 (63.4)
  Change from Baseline to week 52 | -0.5 (11.0) | 0.8 (33.7)

20. Secondary Outcome: Clinical Laboratory Values (Change in Biochemistry - Lactate Dehydrogenase [LDH])
Description: Change from Baseline to Week 52 is calculated from the change in percentage((Week 52 %) - (Baseline %)) per participant, averaged across all participants. Measured in serum at baseline and week 52. Serum samples were analysed at a central laboratory (LDH = lactate dehydrogenase)
Time Frame: Week 0, week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | NN304 | NN729
Number analyzed (Participants) | 164 | 166
U/L
  Baseline | 161.1 (47.8) | 159.4 (57.4)
  Week 52 | 164.9 (62) | 162.7 (37.5)
  Change from Baseline to week 52 | 3.2 (45) | 2.6 (46.7)

21. Secondary Outcome: Clinical Laboratory Values (Change in Biochemistry - Potassium)
Description: as for outcome 11
Time Frame: Week 0, week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | NN304 | NN729
Number analyzed (Participants) | 164 | 166
mmol/L
  Baseline | 4.46 (0.44) | 4.37 (0.49)
  Week 52 | 4.49 (0.49) | 4.43 (0.44)
  Change from Baseline to week 52 | 0.02 (0.50) | 0.06 (0.49)

22. Secondary Outcome: Clinical Laboratory Values (Change in Biochemistry - Sodium)
Description: as for outcome 11
Time Frame: Week 0, week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | NN304 | NN729
Number analyzed (Participants) | 164 | 166
mmol/L
  Baseline | 138.9 (2.6) | 139.2 (2.4)
  Week 52 | 140.3 (2.4) | 140.0 (2.4)
  Change from Baseline to week 52 | 1.4 (2.8) | 0.8 (2.9)

23. Secondary Outcome: Clinical Laboratory Values (Change in Biochemistry - Total Protein)
Description: as for outcome 11
Time Frame: Week 0, week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | NN304 | NN729
Number analyzed (Participants) | 164 | 166
g/dL
  Baseline | 7.23 (0.44) | 7.24 (0.44)
  Week 52 | 7.13 (0.44) | 7.19 (0.43)
  Change from Baseline to week 52 | -0.11 (0.38) | -0.06 (0.37)

24. Secondary Outcome: Adverse Events
Time Frame: Weeks 0-52
Population: as for outcome 1
Measure: Number; unit: events
Arm/Group | NN304 | NN729
Number analyzed (Participants) | 164 | 166
events
  Serious Adverse Events | 25 | 10
  Non-Serious Adverse Events | 259 | 346

ADVERSE EVENTS:
Time Frame: Weeks 0-52
Arm/Group | NN304 | NN729
Serious Adverse Events (participants affected / at risk) | 19/164 | 8/166
Other Adverse Events (participants affected / at risk) | 56/164 | 70/166
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NN304 (N=164) | NN729 (N=166)
Hypoglycaemic Unconsciousness (Metabolism and nutrition disorders) | 3 (4) | 2 (2)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemic (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Ketosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0)
Bronchiectasis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Accidental Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Meniscus Lesion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skull Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bile Duct Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bone Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral Haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Facial Paresis (Nervous system disorders) | 1 (1) | 0 (0)
Hypoglycaemic Coma (Nervous system disorders) | 0 (0) | 1 (1)
Inguinal Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis Relapsing (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lymphadenopathy Mediastinal (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Portal Hypertension (Hepatobiliary disorders) | 0 (0) | 1 (1)
Major Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Vascular Disorders (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NN304 (N=164) | NN729 (N=166)
Nasopharyngitis (Infections and infestations) | 26 (33) | 31 (37)
Influenza (Infections and infestations) | 11 (11) | 11 (17)
Upper Respiratory Tract Infection (Infections and infestations) | 9 (10) | 11 (14)
Headache (Nervous system disorders) | 10 (30) | 17 (59)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
One or more manuscripts for publication will be prepared in collaboration between Investigator(s) and Novo Nordisk. Novo Nordisk will not suppress or veto publications; however Novo Nordisk reserves the right to postpone publication and/or communication for a short time to protect intellectual property.